CLINICAL TRIAL: NCT02913820
Title: Association of Snowfall and Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: EK28-433ex15/16
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- snowfall >5cm/d: impact of snowfall and its correlation with acute myocardial infarctions is analyzed. Other precipitation (rainfall) changes in atmospheric pressure and temperature will be variables to be corrected for.
  Interventions: Other: snowfall > 5cm/day

INTERVENTIONS:
Other: snowfall > 5cm/day — the number of myocardial infarctions of every day analysed in this study will be correlated with the respective values of snowfall

SUMMARY:
Changes in the ambient temperature (esp. warm to cold) as well as exercise are triggers for vasospasms and plaque rupture. Weather data (temperature, precipitation in general as well as snowfall and changes in atmospheric pressure) will be correlated with the incidence of myocardial infarctions.

DETAILED DESCRIPTION:
Besides classical cardiovascular risk factors such as smoking, obesity, elevated cholesterol levels and diabetes there are also acute factors potentially triggering acute coronary events. The impact of air temperature (changes) or humidity are of potential relevance. In addition, exercise and the associated increase in oxygen demand of the myocardium and blood pressure is another trigger for plaque rupture and the acute onset of myocardial infarction. Male patients as well as patients with previous coronary heart disease or little regular exercise are at increased risk.

Possible additional mechanisms of exercise induced myocardial infarction are vasospasm and changes in blood clotting.

Changes in the ambient temperature (warm to cold) can also induce vasospasm which might result in reduced perfusion and plaque rupture. It seems that male patients are more involved than female patients.

Taking the exercise and the ambient temperature changes into consideration, heavy snowfall with consecutive snow shoveling is an augmented risk for acute myocardial infarction.

The rationale of the study is to test if the above mentioned constellation of environmental factors as well as potential increased exercise have a significant and independent impact on the incidence of myocardial infarctions

ELIGIBILITY:
Inclusion Criteria:

* myocardial infarction being confirmed or treated in the cathlab

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with myocardial infarction being transfered to a cath lab either at the medical university of Graz or the department of cardiology at the state hospital Graz West
Sampling Method: Non-Probability Sample
Enrollment: 18075 (Actual)
Dates: Start 2007-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
myocardial infarction | 1 day
  the number of myocardial infarctions of every day analysed in this study will be correlated with the respective values of snowfall

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Result] Burke AP, Farb A, Malcom GT, Liang Y, Smialek JE, Virmani R. Plaque rupture and sudden death related to exertion in men with coronary artery disease. JAMA. 1999 Mar 10;281(10):921-6. doi: 10.1001/jama.281.10.921. PMID 10078489
- [Result] Chevalier L, Hajjar M, Douard H, Cherief A, Dindard JM, Sedze F, Ricard R, Vincent MP, Corneloup L, Gencel L, Carre F. Sports-related acute cardiovascular events in a general population: a French prospective study. Eur J Cardiovasc Prev Rehabil. 2009 Jun;16(3):365-70. doi: 10.1097/HJR.0b013e3283291417. PMID 19318955
- [Result] Gordon JB, Ganz P, Nabel EG, Fish RD, Zebede J, Mudge GH, Alexander RW, Selwyn AP. Atherosclerosis influences the vasomotor response of epicardial coronary arteries to exercise. J Clin Invest. 1989 Jun;83(6):1946-52. doi: 10.1172/JCI114103. PMID 2723067
- [Result] van Teeffelen WM, de Beus MF, Mosterd A, Bots ML, Mosterd WL, Pool J, Doevendans PA, Grobbee DE. Risk factors for exercise-related acute cardiac events. A case-control study. Br J Sports Med. 2009 Sep;43(9):722-5. doi: 10.1136/bjsm.2009.057307. PMID 19734508
- [Result] Willich SN, Lewis M, Lowel H, Arntz HR, Schubert F, Schroder R. Physical exertion as a trigger of acute myocardial infarction. Triggers and Mechanisms of Myocardial Infarction Study Group. N Engl J Med. 1993 Dec 2;329(23):1684-90. doi: 10.1056/NEJM199312023292302. PMID 8232457
- [Result] Giri S, Thompson PD, Kiernan FJ, Clive J, Fram DB, Mitchel JF, Hirst JA, McKay RG, Waters DD. Clinical and angiographic characteristics of exertion-related acute myocardial infarction. JAMA. 1999 Nov 10;282(18):1731-6. doi: 10.1001/jama.282.18.1731. PMID 10568645
- [Result] Ciampricotti R, el Gamal MI, Bonnier JJ, Relik TH. Myocardial infarction and sudden death after sport: acute coronary angiographic findings. Cathet Cardiovasc Diagn. 1989 Aug;17(4):193-7. doi: 10.1002/ccd.1810170402. PMID 2766351
- [Result] Janardhanan R, Henry Z, Hur DJ, Lin CM, Lopez D, Reagan PM, Rudnick SR, Koshko TJ, Keeley EC. The snow-shoveler's ST elevation myocardial infarction. Am J Cardiol. 2010 Aug 15;106(4):596-600. doi: 10.1016/j.amjcard.2010.03.075. PMID 20691323
- [Result] Nitenberg A, Chemla D, Antony I. Epicardial coronary artery constriction to cold pressor test is predictive of cardiovascular events in hypertensive patients with angiographically normal coronary arteries and without other major coronary risk factor. Atherosclerosis. 2004 Mar;173(1):115-23. doi: 10.1016/j.atherosclerosis.2003.12.030. PMID 15177131
- [Result] Thompson DR, Pohl JE, Tse YY, Hiorns RW. Meteorological factors and the time of onset of chest pain in acute myocardial infarction. Int J Biometeorol. 1996 Sep;39(3):116-20. doi: 10.1007/BF01211222. PMID 8937266